CLINICAL TRIAL: NCT03571529
Title: The Effect of EMG-Driven Exoskeleton Robotic Rehabilitation on Improving Hand Functions in Acute Stroke Patients
Brief Title: Robotic Rehabilitation in Patients With Acute Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Collaborators: Medipol University (Other); Medical Park Hospital Istanbul (Other); Rehab-Robotics Company Limited (Industry)
Responsible Party: Principal Investigator, Dilber Karagozoglu Coskunsu, Principal Investigator, Bahçeşehir University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Bahcesehir University
Record Dates: First submitted 2018-04-22; First posted 2018-06-27 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Acute Stroke
Keywords: EMG driven exoskeleton; hand rehabilitation; hand function; upper extremity outcome
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic rehabilitation (Active Comparator): Active Comparator: Robotic rehabilitation
  Protocol with EMG-driven hand exoskeleton (Hand of Hope):
  Warm-up: 10 min passive mode 2 min resting
  Training: According to residual muscle power:
  * 10 min active-assistive, 2 min resting, 10 min Active-assistive or
  * 5 min active, 2 min resting, 15 min active assistive or
  * 10 min active, 2 min resting, 10 min active and
  * 10 min window cleaning game Robotic rehabilitation will be applied 5 times a week; Totally 15 sessions (3 weeks). Conventional physiotherapy also will be performed to the robotic rehabilitation group.
  Interventions: Device: EMG-driven exoskeleton hand robot; Other: Conventional physiotherapy
- conventional physiotherapy (Active Comparator): Conventional Physiotherapy will be performed to the both group 5 sessions a week and totally 15 sessions (3 weeks).
  Conventional physiotherapy will include neurophysiological approaches. Each session will last around 1,5 hours.
  Interventions: Other: Conventional physiotherapy

INTERVENTIONS:
Device: EMG-driven exoskeleton hand robot — Primary Outcome Measurement:
  1. Fugl-Meyer Upper Extremity Assessment
  Secondary Outcome Measurements:
  1. Action Research Arm Test
  2. Motor Activity Log
  3. Data from force and EMG measurement records of HOH robot
  4. Grip strength (with hand dynamometer)
  5. Range of motion measurements of Wrist, and MCP, PIP and DIP joints of the fingers
  6. Manuel muscle testing for wrist and finger muscles.
  7. Modify Asworth sclale At the beginning of each robotic treatment session, superficial EMG recording will be taken at relax position ( without muscle contraction) and then during maximal voluntary isometric contraction (MVC) after the patient's hand is placed in the exoskeleton. For both, EMG recording is performed for 7 seconds and Root Mean Square (RMS) is calculated from this record.
  Arms: Robotic rehabilitation
Other: Conventional physiotherapy — Primary Outcome Measurement:
  1. Fugl-Meyer Upper Extremity Assessment
  Secondary Outcome Measurements:
  1. Action Research Arm Test
  2. Motor Activity Log
  3. Data from force and EMG measurement records of HOH robot
  4. Grip strength (with hand dynamometer)
  5. Range of motion measurements of Wrist, and MCP, PIP and DIP joints of the fingers
  6. Manuel muscle testing for wrist and finger muscles.
  7. Modify Asworth sclale

SUMMARY:
The advantage of the EMG-driven exoskeletons is that patient's own muscle power known as Residual Muscle Power is used to move the extremity while many other robotic devices work and drive impaired limb based on machine directed force. However, it is not clear which group of patients are suitable for EMG driven exoskeletons use and there has not been any established treatment protocol.

The aims of the study are 1- to investigate the effectiveness of the EMG-driven exoskeleton for hand rehabilitation in patients with acute stroke. 2- to understand which group of the patients may give the best response to the EMG-driven technology and how should be the treatment protocol designed.

DETAILED DESCRIPTION:
Improving the rehabilitation outcome of the upper extremity in stroke patients has been an ongoing challenge in the rehabilitation field. Up to 85% of stroke survivors experience a certain degree of paresis of the upper limb at the onset and only 20% to 56% of survivors regain complete functional use of the affected upper limb despite the therapeutic interventions in first 3 months . Recovery of upper limb function is generally slower and non-complete.

To support and speed up a recovery process, there are many robotic devices currently used in the stroke units. Unlike one-on-one treatment applied by clinicans, robotic devices can provide repetitive, task oriented movements,with greater intensity, stimulating and engaging environment for user, hence alleviating the labour-intensive aspects of hands-on conventional therapy. There are a number of complex robotic devices that have been developed over the last two decades to assist upper arm training in rehabilitation.

Using EMG driven exoskeleton, commercially known as the Hand of Hope (HOH), has been shown its efficacy to improve patient's grip and pinch ability, muscle coordination and improve functional daily living tasks in patients even after 3,4,8,10 and 14 years after onset of the stroke. In addition to continuous investigation efforts needed to be spent, there has not been established any treatment protocol using EMG-driven exoskeletons. Since Stroke patients need to be focused on their own residual muscle power, clear indications for EMG-driven exoskeletons i.e., Hand of Hope, need to be established.

An investigation designed to highlight all these points will make an important contribution to the therapeutic approach using EMG-driven hand robotics for the hand rehabilitation after stroke.

ELIGIBILITY:
Inclusion Criteria:

* Having ischemic stroke history within last 4 weeks
* Being at the age 18 and older than 18
* Providing a sitting balance during the robot training (maximum 1 hour with preparation time)
* Understanding and performing simple commands
* Full range of motion in MCP, PIP and DIP
* MAS < 3 for finger flexors and extensors
* Participants who agree to participate in the study

Exclusion Criteria:

* Recurrent stroke
* Other neurologic or orthopedic problems that may affect to upper extremity functions
* Hemispatial neglect (will be diagnosed by Line bisection test and The star cancellation test)
* Refused treatment, non-cooperation
* MAS ≥ 3 (MAS will be measured every week during the treatment period)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-04-06 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Upper Extremity Assessment: | Change from pre-interventional Fugl-Meyer Upper Extremity score at the end of the 15 sessions intervention that will be performed 5 days in a week at a total of 3 weeks.
  Fugl-Meyer assessment was first used in 1975 to assess post-stroke physical performance. 33-item upper extremity subscale of the Fugl-Meyer scale evaluates movements, coordination/speed and pain in the shoulder, elbow, forearm. The highest score for the upper extremity is 66.

SECONDARY OUTCOMES:
Action Research Arm Test (ARAT) | Change from pre-interventional ARAT score at the end of the 15 sessions intervention that will be performed 5 days in a week at a total of 3 weeks.
  ARAT is a performance test, first described by Lyle in 1982. This test is produced by the upper extremity function test and shows upper extremity function and skill. ARAT consists of four subdivisions and 19 functional items that evaluate grasp, grip, pinch and gross motor movement on the both side. The highest score is 57.
Motor Activity Log | Change from pre-interventional Motor Activity Log score at the end of the 15 sessions intervention that will be performed 5 days in a week at a total of 3 weeks.
  Motor Activity Log is a measure used to assess the amount of use and quality of movement of paretic arms and hands in daily living activities for hemiparetic stroke patients. It consists of 30 items.
Manuel muscle testing | Change from pre-interventional Manuel muscle testing scores at the end of the 15 sessions intervention that will be performed 5 days in a week at a total of 3 weeks.
  manuel muscle testing of the flexor and extensor muscles of the wrist and finger
Range of motion measurement (ROM) | Change from pre-interventional ROMs at the end of the 15 sessions intervention that will be performed 5 days in a week at a total of 3 weeks.
  Active range of motion of the wrist, MCP, PIP and DIP joints
Force and EMG measurement with the testing device | Change from pre-interventional force and EMG measurement with the testing device at the end of the 5th session, 10th session and 15 session intervention that will be performed at the last session of each week at a total of 3 weeks.
  Additional force and EMG measurement with the specially designed testing device
hand dynamometer | Change from pre-interventional grip strentgh at the end of the 15 session interventions that will be performed 5 days in a week at a total of 3 weeks.
  to measure grip strength

CONTACTS AND LOCATIONS:
Overall Officials: Dilber Karagozoglu Coskunsu, Ass.Prof., Principal Investigator — Bahçeşehir University; Sumeyye Akcay, PT, Study Chair — Bahçeşehir University; Özden Erkan Oğul, Ass.Prof., Study Chair — Medipol University; Kubra Yıldırım, PT, Study Chair — IAU Medical Park Florya Hospital; Yakup Krespi, Prof., Study Chair — IAU Medical Park Florya Hospital; Haris Begovic, PhD, Study Chair — The Hong Kong Polytechnic University; Necla Öztürk, Prof., Study Chair — Maltepe University
Locations (1):
- Dilber Karagozoglu Coskunsu, Istanbul, Europe, Turkey (Türkiye)